CLINICAL TRIAL: NCT00721591
Title: Pharmacokinetics of Low Molecular Weight and Unfractionated Heparin in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 13677B
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Recurrent Pregnancy Loss; Fetal Demise; Abortion, Habitual; Antiphospholipid Antibodies; Inherited Thrombophilia
Keywords: Recurrent Pregnancy Loss; Habitual abortion; Fetal demise; Antiphospholipid antibodies; Inherited thrombophilia
MeSH Terms: conditions — Fetal Death; Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma from subjects to obtain concentrations of heparin will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Subjects opting for treatment with unfractionated heparin
- B: Subjects opting for treatment with low molecular weight heparin

SUMMARY:
To determine, through pharmacokinetic parameters, the ideal dosing protocol for dalteparin (a low molecular weight heparin) and unfractionated heparin for women desiring pregnancy who have evidence of an acquired (specifically, antiphospholipid syndrome) or inherited thrombophilia.

DETAILED DESCRIPTION:
This study's specific objectives include:

1. Evaluating pharmacokinetic (concentration-time) and pharmacodynamic (concentration- effect) parameters for dalteparin and UFH prior to pregnancy, during the 1st, 2nd and 3rd trimesters and postpartum, using revised dosing protocols based on previous study.
2. Determining therapeutic response to the heparins, i.e. live birth rate and lack of maternal or fetal complications, in relation to drug exposure, based on AUC.
3. Documenting maternal and fetal complications during pregnancy for dalteparin and UFH, using the revised dosing protocols.

ELIGIBILITY:
Inclusion Criteria:

* Two or more consecutive, otherwise unexplained miscarriages under 10 weeks of gestation, or, an otherwise unexplained intrauterine fetal demise of at least 10 weeks of gestation, and,
* Persistently positive antiphospholipid antibodies, or, presence of Factor V Leiden, or, Prothrombin 20210A, or, antithrombin, protein S, or protein C deficiency, or, hyperhomocysteinemia associated with the methylenetetrahydrofolate reductase (MTHFR) polymorphism.

Exclusion Criteria:

* Inability or refusal to give written informed consent.
* Inability or refusal to self-administer heparin throughout pregnancy.
* Hemoglobin value below 9.5 g/dL
* Heparin use is contraindicated.
* Renal disease.
* Documented history of thrombosis.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of 15 subjects prescribed dalteparin and 15 subjects prescribed unfractionated heparin, who are identified through the University of Chicago Recurrent Pregnancy Loss Program.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2005-03; Primary Completion 2013-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The best dosing strategy for either unfractionated or low molecular weight heparin will be the one exhibiting the best balance between a modified Akaike information criterion value, residual sum of squares, and coefficient of determination. | Pre-pregnancy, 1st, 2nd, 3d Trimester and post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Mary D. Stephenson, MD, MSc, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States